CLINICAL TRIAL: NCT00437242
Title: A Study to Evaluate the Effect of Repeat Oral Doses of Odiparcil on Cardiac Conduction as Assessed by 12-lead Electrocardiogram Compared to Placebo and a Single Oral Dose of Moxifloxacin.
Brief Title: Odiparcil QT Definitive Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ITI103221
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Fibrillation, Atrial; Atrial Fibrillation
Keywords: interval,; atrial fibrillation; QT,; odiparcil,
MeSH Terms: conditions — Atrial Fibrillation | interventions — odiparcil

INTERVENTIONS:
Drug: Odiparcil

SUMMARY:
This study is being completed to demonstrate the lack of effect of repeat dosing with Odiparcil on the QTc interval.

ELIGIBILITY:
Inclusion:

* Healthy volunteers

Exclusion:

* Cardiac abnormalities
* Hepatic or renal insufficiency
* Anti-coagulant medications
* Bleeding history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54
Dates: Start 2006-10

PRIMARY OUTCOMES:
demonstrate lack of effect of repeat dose on QT interval with ECG measured on Days -1, 5 and 6 at 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 16, 18, 20 and 24 hours

SECONDARY OUTCOMES:
Pharmacokinetics, CMAX, AUC, TMAX, PK samples taken at 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 16, 18, 20 and 24 hours on days 5 and 6

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States